CLINICAL TRIAL: NCT05192850
Title: Endometrial Cancer Recurrence in Patients Taking Metformin
Status: Withdrawn | Type: Observational
Why Stopped: study was not started at WellSpan
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Eav Lim, Principal Investigator, WellSpan Health
Other Study IDs: 1849612-1
Record Dates: First submitted 2021-12-23; First posted 2022-01-14 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Endometrial Carcinoma
Keywords: metformin; endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Metformin use: These participants were on metformin for any duration at any point in time in the study period
  Interventions: Drug: Metformin use
- No metformin use: These participants were never on metformin for any duration at any point in time in the study period

INTERVENTIONS:
Drug: Metformin use — As an observational study, this is past exposure to metformin that occurred during the study period
  Groups: Metformin use

SUMMARY:
Given the early literature available and its biological plausibility as an inhibitor of the mammalian target of rapamycin (mTOR) protein, it is hypothesized that women with endometrial cancer who take metformin for non-cancer related reasons have a lower cancer recurrence rate compared to women not taking metformin. The primary goal of this study is to determine whether metformin use is associated with a decrease in the rate of endometrial cancer recurrence. Secondary objectives are to assess whether women with endometrial cancer taking metformin have longer progression free survival and overall survival than those that do not take metformin.

DETAILED DESCRIPTION:
This is a retrospective chart review study. Medical records are reviewed and data collected through the hospital's electronic medical record (EMR). Participants are women that had definitive treatment for endometrial cancer between 2016-2020 at WellSpan York Hospital Department of Gynecologic Oncology. Participants are identified and their chart reviewed for demographic data of age, race, comorbid conditions, and use of metformin. Possible confounding information is documented, including chemotherapy status, radiotherapy status, cancer and tumor type, grade, and stage, available genetics information, medications at the time of cancer diagnosis, and medication durations. Those patients who had cancer recurrence are identified. Recurrence data including type, time interval, additional treatment are collected. Recurrence is defined as any recurrence validated by clinical, imaging and histological data and can be identified based on the cancer registry. Recurrence rate in participants that took metformin vs. those that did not is calculated. Time to endometrial cancer recurrence is calculated. Progression free survival and overall survival are calculated. Statistical analysis is performed to compare each of these outcomes between participants who took metformin vs. those that did not.

ELIGIBILITY:
Inclusion Criteria:

* Participants with endometrial cancer of all histologies treated in the WellSpan system from 2016-2020

Exclusion Criteria:

* Participants who underwent palliative treatment for endometrial cancer

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who underwent initial treatment for curative intent of endometrial cancer in the WellSpan system between 2016-2020
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Estimated)

PRIMARY OUTCOMES:
Endometrial Cancer Recurrence | 2016-2020
  This is the identification of whether metformin use is associated with endometrial cancer recurrence.

SECONDARY OUTCOMES:
Progression Free Survival | 2016-2020
  This is the identification of whether metformin use is associated with improved progression free survival of endometrial cancer.
Overall Survival | 2016-2020
  This is the identification of whether metformin use is associated with improved overall survival of endometrial cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Eav Lim, DO, Principal Investigator — WellSpan Health-York Cancer Center
Locations (1):
- WellSpan, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esposito K, Chiodini P, Capuano A, Bellastella G, Maiorino MI, Giugliano D. Metabolic syndrome and endometrial cancer: a meta-analysis. Endocrine. 2014 Feb;45(1):28-36. doi: 10.1007/s12020-013-9973-3. Epub 2013 May 3. PMID 23640372
- [Background] Tang YL, Zhu LY, Li Y, Yu J, Wang J, Zeng XX, Hu KX, Liu JY, Xu JX. Metformin Use Is Associated with Reduced Incidence and Improved Survival of Endometrial Cancer: A Meta-Analysis. Biomed Res Int. 2017;2017:5905384. doi: 10.1155/2017/5905384. Epub 2017 Mar 20. PMID 28409158
- [Background] Tseng CH. Metformin and endometrial cancer risk in Chinese women with type 2 diabetes mellitus in Taiwan. Gynecol Oncol. 2015 Jul;138(1):147-53. doi: 10.1016/j.ygyno.2015.03.059. Epub 2015 Apr 22. PMID 25913129
- [Background] Meireles CG, Pereira SA, Valadares LP, Rego DF, Simeoni LA, Guerra ENS, Lofrano-Porto A. Effects of metformin on endometrial cancer: Systematic review and meta-analysis. Gynecol Oncol. 2017 Oct;147(1):167-180. doi: 10.1016/j.ygyno.2017.07.120. Epub 2017 Jul 29. PMID 28760367
- [Background] Zhang ZJ, Li S. The prognostic value of metformin for cancer patients with concurrent diabetes: a systematic review and meta-analysis. Diabetes Obes Metab. 2014 Aug;16(8):707-10. doi: 10.1111/dom.12267. Epub 2014 Feb 27. PMID 24460896
- [Background] Lee TY, Martinez-Outschoorn UE, Schilder RJ, Kim CH, Richard SD, Rosenblum NG, Johnson JM. Metformin as a Therapeutic Target in Endometrial Cancers. Front Oncol. 2018 Aug 28;8:341. doi: 10.3389/fonc.2018.00341. eCollection 2018. PMID 30211120
- [Background] Xie W, Li T, Yang J, Shang M, Xiao Y, Li Q, Yang J. Metformin use and survival outcomes in endometrial cancer: a systematic review and meta-analysis. Oncotarget. 2017 Aug 22;8(42):73079-73086. doi: 10.18632/oncotarget.20388. eCollection 2017 Sep 22. PMID 29069850